CLINICAL TRIAL: NCT02324296
Title: PEI REGIMEN: A THERAPEUTIC OPTION IN SMALL CELL LUNG CANCER? A MONOINSTITUTIONAL EXPERIENCE OF 46 CONSECUTIVE CASES
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: PEI 01
Record Dates: First submitted 2014-12-11; First posted 2014-12-24 (Estimated); Last update posted 2025-06-11 (Actual); Status verified 2014-12

CONDITIONS: Small Cell Lung Cancer
Keywords: small cell lung cancer; extended disease; limited disease; chemotherapy; cisplatin; etoposide; ifosfamide
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Ifosfamide; PE regimen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ifosfamide — PEI regimen may be a possible therapeutic option, with high activity and an acceptable toxicity profile.
  Other Names: cisplatin, etoposide

SUMMARY:
ABSTRACT Objectives Combination chemotherapy is very active in small cell lung cancer (SCLC), although no improvement in overall survival (OS) has been done in the last 25 years , with Cisplatin-Etoposide (PE) still considered the world-wide standard, with an average median survival of about 7-8 months in patients with extended disease (ED).

In 1995, a randomized trial of the Hoosier Group in 171 ED patients showed a significant advantage in overall survival in patients treated with PEI (Cisplatin, Etoposide and Ifosfamide), compared to PE. Despite that, PEI regimen has not become a commonly used regimen in SCLC.

Materials and Methods Here we present a series of 46 consecutive patients (30 males and 16 females) with SCLC that were treated at our Institution with PEI regimen: Cisplatin 20mg/m2, Etoposide 75mg/m2 and Ifosfamide 1200mg/m2, day 1 to 4, every 3 weeks.

Patients received a total of 219 cycles of chemotherapy, with a mean of 4,7 cycles per patient. Median age was 63 (range 59-70); performance status (PS) was 0 in 29 patients (63%), 1 in 13 patients (28%) and 2 in 4 patients (9%).

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically proven SCLC
* measurable disease defined by RECIST criteria

Exclusion Criteria:

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients had histologically or cytologically proven SCLC, with measurable disease defined by RECIST criteria, and received at least one cycle of chemotherapy. Patients with central nervous system (CNS) metastases were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 1998-12; Primary Completion 2009-01 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
partial response (PR) | 1 year
complete response (CR) | 1 YEAR

SECONDARY OUTCOMES:
Median time to progression (TTP) | 1 YEAR
overall survival (OS) | 1 YEAR

REFERENCES:
- [Derived] Boni C, Pagano M, Baldi L, Gnoni R, Braglia L, Savoldi L, Zanelli F. Pei regimen: a therapeutic option in small cell lung cancer? A retrospective monoinstitutional analysis of 46 consecutive cases. J Transl Med. 2015 Apr 24;13:130. doi: 10.1186/s12967-015-0491-3. PMID 25903963